CLINICAL TRIAL: NCT02845869
Title: Evaluation of the Efficacy of Light Therapy for the Treatment of Anterior Knee Pain: A Prospective, Randomized, Double-Blind, Sham-Controlled Clinical Trial
Brief Title: Evaluating Light Therapy for Treatment of Overuse Anterior Knee Pain
Acronym: LLL&KP02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Shaare Zedek Medical Center (Other); International Diabetes Federation (Other)
Responsible Party: Principal Investigator, Lilach Gavish, Study Director, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0130-16-SZMC
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light Therapy (Experimental): Subjects from this group will receive 8 biweekly physiotherapy treatment and in addition Light Therapy treatment with the THOR laser LX2 system.
  Interventions: Device: THOR Laser LX2 System
- Sham Therapy (Sham Comparator): Subjects from this group will receive 8 biweekly physiotherapy treatment and in addition Sham Therapy.
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: THOR Laser LX2 System — Treatment session will take up to 25 minutes and will include stimulation of local lymph nodes and soft tissue, de-activation of trigger points, and eliciting analgesia.
  Arms: Light Therapy
Device: Sham Therapy — The therapeutic light will be turned off but the system will produce similar noises and mild heat.
  Arms: Sham Therapy

SUMMARY:
During basic training, 15% of military recruits develop knee pain, which hinders their chance to complete training. Current therapeutic options have had variable levels of success. Light therapy was shown to reduce pain in chronic inflammatory related knee pathology. The current clinical study is designed to evaluate light therapy, as an adjunct to conservative physiotherapy for treatment of acute overuse KP in combat soldiers.

DETAILED DESCRIPTION:
During basic training, 15% of military recruits develop knee pain on the background of overuse, which hinders their chance to complete training, and leads to high dropout rate with the accompanying cost to the system. When KP is due to overuse, the time to complete resolution is typically 2-3 months, but symptoms may last for years. Current therapeutic options have had variable levels of success. Finding an alternative non-drug, non-invasive therapeutic modality that is easily incorporated in a field setting and may shorten the resolution of pain may lead to earlier return to duty thereby reducing the associated cost to the system and to the individual soldier.

Low-level laser irradiation (LLLI) is non-ionizing and non-thermal, and is within the visible to near-infrared range of the electromagnetic spectrum. LLLI has been used widely for alleviation of pain, reduction of inflammation, and acceleration of wound healing. Pre-clinical and clinical studies have shown that LLLI reduces pain in chronic inflammatory related knee pathology. However, little is known about the effect of LLLI on acute knee pathology that account for 25-40% of all knee problems in athletes.

The current study is a prospective, randomized, controlled double blind clinical study designed to evaluate light therapy, as an adjunct to conservative physiotherapy for treatment of acute overuse KP in combat soldiers.

The treatment protocol includes conservative physiotherapy and in addition, biweekly sessions of light therapy or sham irradiation for 4 weeks. Two follow up visits will take place at 1 week and 3 months after the last treatment.

Study evaluations will include physical examination, physical activity tests, subjective pain level by visual analogue scale, improvement and satisfaction scores, and functional questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 65
2. Knee pain on the background of overuse as determined by the orthopedic surgeon
3. Willing to sign informed consent

Exclusion Criteria:

1. Previous trauma to the knee
2. Previous or planned surgical treatment to the knee
3. Suspected meniscus injury
4. Suffering from significant concurrent illness, such as cardiac disorders, or pertinent neurological disorders.
5. Suffering from condition that does not permit filling questionnaires
6. Use of NSAIDs during the 2 weeks before the development of Knee pain or before receiving treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatments in subjective pain level using a Visual Analogue Scale (VAS) | 1 month (end of treatments)
  Subject assessment of pain will be evaluated using a Visual Analogue Scale (VAS), were 0 is "no pain" and 100 is "intolerable pain"

SECONDARY OUTCOMES:
Change from baseline to 3 month follow up in subjective pain level using a Visual Analogue Scale (VAS) | 3 month post treatments
  Subject assessment of pain will be evaluated using a Visual Analogue Scale (VAS), were 0 is "no pain" and 100 is "intolerable pain"

CONTACTS AND LOCATIONS:
Overall Officials: Yair Barzilay, MD, Principal Investigator — Shaare Zedek Hospital; Lilach Gavish, PhD, Study Director — HUJI
Locations (1):
- IDF bases, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gavish L, Spitzer E, Friedman I, Lowe J, Folk N, Zarbiv Y, Gelman E, Vishnevski L, Fatale E, Herman M, Gofshtein R, Gam A, Gertz SD, Eisenkraft A, Barzilay Y. Photobiomodulation as an Adjunctive Treatment to Physiotherapy for Reduction of Anterior Knee Pain in Combat Soldiers: A Prospective, Double-Blind, Randomized, Pragmatic, Sham-Controlled Trial. Lasers Surg Med. 2021 Dec;53(10):1376-1385. doi: 10.1002/lsm.23442. Epub 2021 Jun 8. PMID 34101208